CLINICAL TRIAL: NCT06981819
Title: Establishment and Effectiveness Evaluation of a Training System for Confocal Laser Endomicroscopy in Diagnosing Gastric Neoplastic Lesions: A Prospective Diagnostic Study
Brief Title: Establishment and Effectiveness Evaluation of a Training System for Confocal Laser Endomicroscopy
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: China Biotechnology Development Center (Unknown)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: CLE Training
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Gastric High-grade Intraepithelial Neoplasia; Gastric Low-grade Intraepithelial Neoplasia; Gastritis
Keywords: Confocal Laser Endomicroscopy; Gastric Neoplastic Lesions
MeSH Terms: conditions — Stomach Neoplasms; Gastritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric mucosal biopsy specimens or resected specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Probe-based Confocal Laser Endomicroscopy by Experts — Confocal Laser Endomicroscopy (CLE) is an advanced in vivo imaging technique that combines confocal microscopy with endoscopy, enabling real-time, microscopic visualization of tissues at a cellular level during endoscopic procedures. Probe-based CLE (pCLE) can enter the stomach cavity through the biopsy channel of the endoscope and observe the gastric mucosa. To generate diagnostic results of pCLE, two pCLE experts dignosed independent. Any discrepancies are then resolved by a third expert.
  Other Names: pCLE by Experts
Diagnostic Test: magnifying endoscopy with blue laser imaging — Magnifying Endoscopy with Blue Laser Imaging (ME-BLI) is an advanced endoscopic imaging technique that combines high-resolution magnification with laser-enhanced visualization to improve the detection and characterization of gastrointestinal (GI) mucosal lesions. Developed by Fujifilm, BLI utilizes specific laser wavelengths to enhance surface and vascular patterns, making it particularly useful for diagnosing early-stage cancers and precancerous conditions in the stomach, colon, and esophagus. To generate diagnostic results of ME-BLI, two ME-BLI experts dignosed independent. Any discrepancies are then resolved by a third expert.
  Other Names: ME-BLI
Diagnostic Test: Probe-based Confocal Laser Endomicroscopy by trainees — Confocal Laser Endomicroscopy (CLE) is an advanced in vivo imaging technique that combines confocal microscopy with endoscopy, enabling real-time, microscopic visualization of tissues at a cellular level during endoscopic procedures. Probe-based CLE (pCLE) can enter the stomach cavity through the biopsy channel of the endoscope and observe the gastric mucosa. The diagnosis results of CLE trainees are generated by each trainee themselves.
  Other Names: pCLE by trainees

SUMMARY:
Gastrointestinal endoscopy is a vital method for screening and diagnosing gastric cancer. It aids in identifying the tumor's location within the stomach and its macroscopic type, and allows biopsy for histological confirmation. Moreover, suspicious lesions can be further examined using specialized endoscopic techniques such as magnifying endoscopy (ME) combined with electronic staining, chromoendoscopy, confocal laser endomicroscopy (CLE) and fluorescence endoscopy. ME combined with electronic staining has been confirmed to achieve excellent diagnostic accuracy in distinguishing between noncancerous and cancerous lesions. However, ME is technically challenging, and gastric magnifying endoscopy involves various evaluation criteria such as the vessel plus surface classification system and Kudo's pit pattern classification, leading to a steep learning curve.

Confocal Laser Endomicroscopy (CLE) is an advanced in vivo imaging technique that combines confocal microscopy with endoscopy, enabling real-time, microscopic visualization of tissues at a cellular level during endoscopic procedures. Despite having been available for approximately 20 years, and its accuracy in diagnosing gastric neoplastic lesions having been confirmed by several studies, the clinical application of CLE is not widespread, and there is a lack of relevant standards to guide the training of CLE endoscopists. To train more CLE endoscopists, we organized CLE training courses. We also evaluated the training's effectiveness and try to explore the Influencing factors of learning curve.

ELIGIBILITY:
Inclusion Criteria:

* atients aged 18 to 85 years who were scheduled for detailed endoscopic examination at the First Affiliated Hospital of Naval Medical University were consecutively enrolled.

Exclusion Criteria:

* nwillingness to undergo CLE examination
* hypersensitivity to sodium fluorescein
* hepatic or renal insufficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The use of detailed endoscopic examination includes the following scenarios: routine endoscopic examination suspected early cancer but the biopsy pathology only indicated precancerous lesions, preoperative examination for early upper gastrointestinal cancer endoscopic resection, follow-up after endoscopic resection of early upper gastrointestinal cancer and precancerous lesions, follow-up after partial gastrectomy for advanced gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | From enrollment to obtaining the pathological results at 2 weeks
  Diagnostic accuracy in the research refers to the ability of diagnostic tests to correctly identify gastric cancerous or noncancerous lesions. gastric cancerous lesions included gastric high-grade intraepithelial neoplasia (HGIN), and gastric cancer. The calculation method for diagnostic accuracy is the percentage of cases where the diagnostic results are consistent with the pathological results out of the total number of cases.

SECONDARY OUTCOMES:
Other diagnostic performance outcomes | From enrollment to obtaining the pathological results at 2 weeks
  Other diagnostic performance outcomes included diagnostic sensitivity, specificity, positive predictive value and negative predictive value.
Kappa value | From the completion of the diagnosis of all cases to the end of calculating the Kapper value at one week.
  The Kappa value was used to evaluate the reliability or agreement between two diagnostic methods or two diagnostic results. In this study, the pathological results were used as the gold standard. The pCLE diagnosis results of each trainee were compared for consistency with the expert's pCLE results as well as the expert's ME-BLI diagnosis results using the Kapper value. The pCLE results and the ME-BLI diagnosis results provided by the experts also need to be compared for consistency using the Kapper value.

OTHER OUTCOMES:
Influencing factors of learning curve of pCLE | From the complete the diagnosis by all the trainees to completion the factor analysis at 2 weeks
  We try to explore the Influencing factors of learning curve of pCLE in this research. To investigate factors that might influence the learning curve of pCLE, several factors were taken into account, including professional title, hospital level, number of endoscopic cases, number of ME cases, and duration of ME usage.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Naval Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided